CLINICAL TRIAL: NCT03429218
Title: A Phase I, First-in-human, Open-label, Dose-escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Oral TP-0184 Administered Once Weekly for 4 Weeks to Patients With Advanced Solid Tumors
Brief Title: First-in-human Study of Oral TP-0184 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0184-101
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumors
Keywords: Sumitomo Dainippon Pharma Oncology SDPO; Phase 1; First in human; Solid Tumors; Advanced Malignancy; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm TP-0184 (Experimental): Weekly dose of TP-0184 by oral administration
  Interventions: Drug: TP-0184

INTERVENTIONS:
Drug: TP-0184 — Oral dose once weekly for 4 weeks

SUMMARY:
TP-0184 is a potent inhibitor of ALK2 or ACRV1 kinase, a constitutively active serine/threonine receptor kinase due to activating mutations or upregulated upstream signaling pathways. This is a Phase 1, open-label, dose-escalation, safety, pharmacokinetics, and pharmacodynamic study, with a purpose of determining the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of oral TP-0184 administered once weekly for 4 weeks in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs) of oral TP-0184 administered once weekly for 4 weeks, over a range of doses in patients with advanced solid tumors.

Secondary Objectives:

* To establish the pharmacokinetics of orally administered TP-0184
* To observe patients for any evidence of antitumor activity of TP-0184 by objective radiographic assessment
* To study the pharmacodynamics of TP-0184 therapy
* To establish the Recommended Phase 2 Dose (RP2D) for future studies with TP-0184

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically confirmed diagnosis of advanced metastatic or progressive solid tumor
2. Be refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition.
3. Have one or more tumors measurable or evaluable as outlined by modified RECIST v1.1
4. Have an Eastern Cooperative Oncology Group (ECOG) (World Health Organization [WHO]) performance of ≤1
5. Have a life expectancy ≥3 months
6. Be ≥18 years of age
7. Have a negative pregnancy test (if female of childbearing potential)
8. Have acceptable liver function:

   1. Bilirubin ≤1.5x upper limit of normal (ULN)
   2. Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) and alkaline phosphatase ≤2.5x upper limit of normal (ULN) *If liver metastases are present, then ≤5x ULN is allowed.
9. Have acceptable renal function: Calculated creatinine clearance ≥ 30 mL/min
10. Have acceptable hematologic status:

    1. Granulocyte ≥1500 cells/mm3
    2. Platelet count ≥100,000 (plt/mm3)
    3. Hemoglobin ≥8 g/dL (Patients may not have received prior transfusions within 2 weeks of the first dose of TP-0184)
11. Have acceptable coagulation status:

    1. Prothrombin time (PT) within 1.5x normal limits
    2. Activated partial thromboplastin time (aPTT) within 1.5x normal limits
12. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an effective method of contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation and for at least 3 months (males) and 6 months (females) after the last study drug dose. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
13. Have read and signed the Institutional Review Board (IRB)-approved informed consent form (ICF) prior to any study related procedure. (In the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new ICF must be signed.)

Exclusion Criteria:

1. History of congestive heart failure (CHF); cardiac disease, myocardial infarction within the past 6 months prior to Cycle 1 Day 1; left ventricular ejection fraction (LVEF) <45% by echocardiogram (ECHO), unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG) within 14 days prior to Cycle 1 Day 1
2. Have a corrected QT interval (using Fridericia's correction formula) (QTcF) of >450 msec in men and >470 msec in women
3. Have a seizure disorder requiring anticonvulsant therapy
4. Presence of symptomatic central nervous system metastatic disease or disease that requires local therapy such as radiotherapy, surgery, or increasing dose of steroids within the prior 2 weeks
5. Have severe chronic obstructive pulmonary disease with hypoxemia (defined as resting O2 saturation of ≤90% breathing room air)
6. Have undergone major surgery, other than diagnostic surgery, within 2 weeks prior to Cycle 1 Day 1
7. Have active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
8. Are pregnant or nursing
9. Received treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 28 days or 5 half lives, whichever occurs first, prior to study entry (6 weeks for nitrosoureas or Mitomycin C)
10. Are unwilling or unable to comply with procedures required in this protocol
11. Have known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. Patients with history of chronic hepatitis that is currently not active are eligible.
12. Have a serious nonmalignant disease (eg, hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
13. Are currently receiving any other investigational agent
14. Have exhibited allergic reactions to a similar structural compound, biological agent, or formulation
15. Have undergone significant surgery to the gastrointestinal tract that could impair absorption or that could result in short bowel syndrome with diarrhea due to malabsorption
16. Have hemochromatosis or a transferrin saturation (TS) >50% in men or >45% in women at baseline or noted during the study via scheduled iron panel monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) and treatment emergent adverse events | Day 1 - 28
  A DLT is defined as any one of the following events observed within Cycle 1 regardless of investigator attribution unless there is a clear alternative explanation:
  * Grade 3 or greater febrile neutropenia
  * Grade 4 neutropenia for ≥7 consecutive days
  * Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with clinically significant bleeding or that requires a platelet transfusion
  * Grade 3 or 4 nonhematologic AEs including nausea, vomiting, diarrhea, and electrolyte imbalances persisting for more than 48 hours despite optimal medical management
  * Dosing delays ≥1 week due to treatment emergent adverse events or related severe laboratory test values
Determine maximum tolerated dose (MTD) | 20 months
  If a patient experiences a DLT, up to three additional patients will be treated at that dose level. If no additional DLTs are observed in the expanded six-patient cohort, the dose will be escalated in a new cohort of three patients. If two or more patients at a given dose level experience a DLT during the first cycle, then the MTD will have been exceeded and up to a total of six patients will be treated at the next lower dose level. If 0 or 1 of 6 patients experiences a DLT at this previous lower dose level, this dose will be declared the MTD.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose of TP-0184 | 23 months
  To establish the Recommended Phase 2 Dose (RP2D) for future studies with TP-0184, MTD data to be reviewed
Determine antitumor activity of TP-0184 | 20 months
  Objective radiographic assessment to be performed to determine antitumor activity by modified RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Greg Pennock, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (5):
- United States (5):
  - Honor Health, Scottsdale, Arizona
  - Northside Hospital, Atlanta, Georgia
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Massachusetts General Hospital MGH, Boston, Massachusetts
  - University of Texas Southwestern UTSW, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No